CLINICAL TRIAL: NCT03802045
Title: Electroacupuncture Frequency-related Effects on Chronic Low Back Pain in Older Adults: Triple-blind, 12-month Protocol for a Randomized Controlled Trial.
Brief Title: Electroacupuncture Frequency-related Effects on Non-specific Low Back Pain in Older Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USaoPauloSA
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Low Back Pain
Keywords: Acupuncture; Electroacupuncture; Low back pain; Aged; Clinical trial
MeSH Terms: conditions — Low Back Pain | interventions — Electroacupuncture; Acupuncture Therapy; Needles

STUDY DESIGN:
Intervention Model Description: The individuals will be randomly assigned to one of five treatment groups: Low frequency EA (LF) with 2Hz, high frequency EA (HF) with 100Hz, alternating frequency EA (AF) with 2 and 100Hz for 3 seconds each, control group (C) and placebo group (P), each containing 25 participants. The LF, HF and AF groups will be submitted to the treatment protocol, which will consist of the bilateral application of electroacupuncture using NKL® portable electrostimulator. The C and P groups will follow exactly the same protocol as the electroacupuncture groups, however the C group will not undergo electrical stimulation, as the acupuncturist will activate channels that are not connected to the patient. In the P group an adhesive moxa will be placed on each acupoint and the needle will be inserted over it. In addition, as in group C, the electrodes will be connected to the needles, however, no electrical current will be applied.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Prior to the first treatment session, the random allocation sequence will be implemented by a researcher not involved in the patient recruitment or evaluation, and will be generated through the randomization.com program, where each number will match one of five study groups.
  After the numbers are generated, they will be placed in sealed, brown envelopes and numbered in series, then given to the acupuncturist. This person will open them according to the numerical sequence, prior to the first session.
  Patients will remain blind regarding the category of their allocation throughout the data collection period of the study. Additionally, the evaluators responsible for the data collection and the outcomes assessor will be blinded to the patient allocation. The acupuncturist, being responsible for the interventions, will be the only person not blind to the type of treatment to be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Low frequency EA (Experimental): 25 participants will receive bilateral application of electroacupuncture using a previously calibrated EL 608 electrostimulator (NKL® portable), with the following parameters: balanced asymmetrical biphasic polarized pulse with continuous pulse train with 2Hz; 100ms pulse duration and 0.5ms pulse width; and the maximum current (amplitude) intensity tolerated by the patient and intensified so that sensory habituation is avoided. Trichotomy will be carried out when necessary and the skin will be disinfected with 70% alcohol. With the participant lying down in a ventral position, the needles will be inserted at a 90º inclination with the skin, to a depth at which that the patient reports the "deQi" sensation (≅ 1.5cm).
  Interventions: Procedure: Electroacupuncture; Device: Needle
- High frequency EA (Experimental): 25 participants will receive 25 participants will receive bilateral application of electroacupuncture using a previously calibrated EL 608 electrostimulator (NKL® portable), with the following parameters: balanced asymmetrical biphasic polarized pulse with continuous pulse train with 100Hz; 100ms pulse duration and 0.5ms pulse width; and the maximum current (amplitude) intensity tolerated by the patient and intensified so that sensory habituation is avoided. Trichotomy will be carried out when necessary and the skin will be disinfected with 70% alcohol. With the participant lying down in a ventral position, the needles will be inserted at a 90º inclination with the skin, to a depth at which that the patient reports the "deQi" sensation (≅ 1.5cm).
  Sterile and disposable 0.25mm x 30mm stainless steel needles (Dong Bang Acupuncture Inc., Seoul, Korea) will be used. The sessions will last 30 minutes, twice a week, for 5 weeks, totaling 10 sessions.
  Interventions: Procedure: Electroacupuncture; Device: Needle
- Alternating frequency EA (Experimental): 25 participants will receive 25 participants will receive bilateral application of electroacupuncture using a previously calibrated EL 608 electrostimulator (NKL® portable), with the following parameters: balanced asymmetrical biphasic polarized pulse with continuous pulse train with 100Hz and 2Hz for 3 seconds each; 100ms pulse duration and 0.5ms pulse width; and the maximum current (amplitude) intensity tolerated by the patient and intensified so that sensory habituation is avoided. Trichotomy will be carried out when necessary and the skin will be disinfected with 70% alcohol. With the participant lying down in a ventral position, the needles will be inserted at a 90º inclination with the skin, to a depth at which that the patient reports the "deQi" sensation (≅ 1.5cm).
  Sterile and disposable 0.25mm x 30mm stainless steel needles (Dong Bang Acupuncture Inc., Seoul, Korea) will be used. The sessions will last 30 minutes, twice a week, for 5 weeks, totaling 10 sessions.
  Interventions: Procedure: Electroacupuncture; Device: Needle
- Control Group (Active Comparator): 25 participants will follow exactly the same protocol as the experimental groups, however they will not undergo electrical stimulation, as the acupuncturist will activate channels that are not connected to the patient.
  Sterile and disposable 0.25mm x 30mm stainless steel needles (Dong Bang Acupuncture Inc., Seoul, Korea) will be used. The sessions will last 30 minutes, twice a week, for 5 weeks, totaling 10 sessions.
  Interventions: Device: Needle
- Placebo Group (Placebo Comparator): 25 participants will will follow exactly the same protocol as the experimental groups, however an adhesive moxa (Dong Yang®) will be placed on each acupoint and the needle will be inserted over it, so that the participant only feels the needle prick, but without perforation of the skin and the "deQi" sensation. In addition, as in the control group, the electrodes will be connected to the needles, however, no electrical current will be applied.
  Sterile and disposable 0.25mm x 30mm stainless steel needles (Dong Bang Acupuncture Inc., Seoul, Korea) will be used. The sessions will last 30 minutes, twice a week, for 5 weeks, totaling 10 sessions.
  Interventions: Device: Needle; Device: Adhesive Moxa

INTERVENTIONS:
Procedure: Electroacupuncture — The interventions will be performed by acupuncture specialists with at least 3 years of clinical experience, who will receive prior training to ensure that they rigorously follow the study protocol and are familiar with the types of treatments, including details such as acupuncture points and manipulation of electroacupuncture parameters.
  After the randomization, the acupuncturist will sequentially open the envelopes, and the individuals will be randomly assigned to one of five treatment groups: Low frequency EA (LF), high frequency EA (HF), alternating frequency EA (AF), control group (C) and placebo group (P), each containing 25 participants. The acupuncture points will be located and described according to the WHO Standard Acupuncture Locations. Based on the beneficial effects of previous clinical trials, the acupoints selected for this study will be: BL23, BL25, BL40, SP6 and KI3.
  Other Names: Acupuncture
  Arms: Alternating frequency EA; High frequency EA; Low frequency EA
Device: Needle — Sterile and disposable 0.25mm x 30mm stainless steel needles (Dong Bang Acupuncture Inc., Seoul, Korea) will be used.
Device: Adhesive Moxa — In the placebo group an adhesive moxa will be placed on each acupoint and the needle will be inserted over it.
  Arms: Placebo Group

SUMMARY:
Background: Low back pain (LBP) is the most frequent complaint in the clinical practice. Electroacupuncture treatment may be effective, however, the evidence supporting this possibility is still limited, especially in older adults.

Methods: A five-arm randomized controlled trial with patients and evaluators blinded to the group allocation. A total of 125 participants with non-specific low back pain will be randomly assigned into one of five groups: three electroacupuncture groups (low, high and alternating frequency), a control and a placebo group. The electroacupuncture will be applied twice a week (30 minutes per session) for 5 weeks. The primary clinical outcome will be pain intensity. The secondary outcomes include: quality of pain, physical functioning, perceived overall effect, emotional functionality, patient satisfaction and psychosocial factors. Patients will be evaluated before the first session, immediately after the last, and followed-up after 6 and 12 months to check the effects in the medium and long term.

Discussion: Results of this trial will help clarify the therapeutic effect of different frequencies of electroacupuncture for chronic low back pain in older adults and to determine the most effective electroacupuncture frequency.

DETAILED DESCRIPTION:
This study will be a randomized controlled clinical trial with blind evaluators and patients. The study will be conducted at the University of São Paulo (USP), approved by the Research Ethics Committee of the Medical School of USP (authorization No. 2.903.991) and financed with its own resources.

Participants will be recruited through radio ads, social networks and local newspapers. Individuals will be informed about the research proposal and treatment protocol, and those that are interested in participating will be selected according to the inclusion and exclusion criteria.

Patients will be eligible for inclusion if they are over 60 years of age, of either gender, with diagnosis of nonspecific LBP of more than 3 months duration, with or without radiating leg pain, with a minimum pain intensity score of 4 on the 11-point pain numerical rating scale (NRS - Brazilian Portuguese version), that can walk independently (with or without walking devices) and that agree to voluntarily participate in this study and sign the consent form.

Patients will be excluded if they have had previous surgery on the spinal column, have a known or suspected serious spinal pathology (e.g., cancer, vertebral fracture, spinal infection or cauda equina syndrome), a fear of needles, have participated in acupuncture treatment in the previous 30 days, if they are wheelchair users, or if they are unable to sign the consent form.

The protocol of this study is based on standards established under the Standards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA) and the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT).

Prior to the first treatment session, the random allocation sequence will be implemented by a researcher not involved in the patient recruitment or evaluation, and will be generated through the randomization.com program, where each number will match one of five study groups.

After the numbers are generated, they will be placed in sealed, brown envelopes and numbered in series, then given to the acupuncturist. This person will open them according to the numerical sequence, prior to the first session.

Patients will remain blind regarding the category of their allocation throughout the data collection period of the study. Additionally, the evaluators responsible for the data collection will be blinded to the patient allocation. The acupuncturist, being responsible for the interventions, will be the only person not blind to the type of treatment to be performed.

The interventions will be performed by acupuncture specialists with at least 3 years of clinical experience, who will receive prior training to ensure that they rigorously follow the study protocol and are familiar with the types of treatments, including details such as acupuncture points and manipulation of electroacupuncture parameters.

Outcome measures Four stages of evaluations will be performed: prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment. The evaluators will be trained in advance.

The primary clinical outcome will be pain intensity. The secondary outcomes will include quality of pain, physical functioning, perception of overall effect, emotional functionality, patient satisfaction and psychosocial factors. All the scales and questionnaires have been translated into Brazilian Portuguese, with the exception of the visual analog scale for the assessment of anxiety, and their properties clinimetrically tested.

Primary outcomes Pain intensity Numerical Rating Scale (NRS) The NRS is an 11-point scale ranging from 0 (no pain) to 10 (worst possible pain). Participants will be asked to rate their average pain levels in the 24 hours prior to the assessment.

Pressure pain threshold (PPT) The pressure pain threshold (PPT) will be measured using a pressure algometer (EMG system, Brazil). The assessed region will be marked with a tape measure and a dermatographic pencil. Two points will be marked bilaterally: 5 cm to the right and left of the spinous process of L3 and L5. A control point will be marked on the anterior tibial muscle of the right leg, 5 cm lateral to the tuberosity of the tibia. The circular tip of the algometer will be positioned perpendicular to the participant's skin and gradually pressed until the participant reports that the pressure has become painful and unbearable. Three measurements will be taken at each point with an interval of 1 minute. At the end, the arithmetic mean will be used to define the pressure pain threshold. To ensure data reliability, a preliminary intra-observer study will be conducted to measure the pressure pain threshold at the assessment points that will be used in the study. In this, 10 participants will be evaluated and reassessed by the same examiner, with a 48-hour interval. The intraclass correlation coefficient (ICC) will be calculated by the measurements of the PPT of the anterior tibial and the lumbar points.

Secondary outcomes Quality of pain This will be analyzed using the McGill Pain Questionnaire, a valid and reliable instrument containing 78 pain descriptors divided into 4 categories (sensory, affective, evaluative and miscellaneous) and 20 subcategories, to which scores of 1 to 5 are attributed. The result is obtained by first scoring the words according to their position within the set of descriptors of each subcategory. The maximum score in the sensory category is 42, in the affective 14, in the evaluative 5 and in the miscellaneous 17. Then, the analysis is performed by adding these values associated with their categories. Higher scores equate to more intense pain. Physical functioning This measure will be assessed through the Roland Morris Disability Questionnaire and the Five Times Sit to Stand Test (FTSST).

The first is a self-administered questionnaire, adapted to the Portuguese language, which aims to evaluate physical incapacity due to low back pain. This contains 24 items pertaining to activities that can be impaired due to LBP. Individuals need to select the items that apply to their pain on that day. The selected items are summed for a total score ranging from 0 to 24, with higher scores indicating more severe functional incapacity. The activity of sitting and standing is a common and important movement in daily life, and in the clinical practice it helps to determine a person's functional level. The patient initiates the FTSST sitting in a chair without arm support, with the upper limbs crossed over the chest, feet positioned at hip width and knees in 90° flexion. They will be asked to stand and sit five times as fast as possible. A timer will be used to measure the task execution time. The test will be performed twice and the mean time will be calculated.

Perceived overall effect The patient's self-perception regarding the treatment will be evaluated using the Global Effect Perception Scale, a 11-point numerical scale ranging from -5 (much worse) to +5 (much better), where higher scores represent better recovery.(18) Emotional functionality Depression and anxiety will be assessed using the Beck Depression Inventory (BDI) and the Global Anxiety - Visual Analog Scale (GA-VAS), respectively.

The BDI is a self-administered questionnaire that contains 21 items, with a score ranging from 0 to 3, where a higher score indicates more depressive symptoms. The GA-VAS is composed of a 100mm line, where the left extremity is related to the absence of anxiety, and the right extremity is related to the worst possible anxiety. The individual is asked to assess the intensity of their anxiety in the previous 24 hours and to mark this on the line. The distance from the left edge of the line to the mark placed by the patient is measured in millimeters. Greater measurements indicate greater anxiety.

Patient satisfaction The evaluation of the patient's satisfaction with the treatment will be carried out using the MedRisk questionnaire of patient satisfaction with physiotherapeutic care. This questionnaire contains 20 items, covering global aspects of the treatment (2 items), aspects related to the service provided (8 items), and aspects about the therapist-patient relationship (10 items). Following a Likert-type scale, the patient's response will range from 1 (strongly disagree) to 5 (strongly agree), where higher scores represent greater satisfaction with the treatment.

Psychosocial factors The risk of a poor prognosis due to psychosocial factors will be assessed using the STarT Back Screening Tool (SBST), a self-administered questionnaire with 9 items (4 related to referred pain and 5 related to psychosocial factors) where the patient has the response options "I agree" (1 point) and "I Disagree" (zero points) in the first eight items, and "Nothing", "A little" or "Moderate" (zero points each), "A lot" or "Extremely" (one point each) in the ninth item. If the total score is between 0-3 points, the patient is classified as low risk for poor prognosis. When the total score is greater than 3 points the score of the psychosocial subscale, questions 5 to 9, is then considered. If the score of this subscale is less than or equal to 3 points, the patient is classified as medium risk and scores greater than 3 points are considered to indicate a high risk for poor prognosis. Procedures After the randomization, the acupuncturist will sequentially open the envelopes, and the individuals will be randomly assigned to one of five treatment groups: Low frequency EA (LF), high frequency EA (HF), alternating frequency EA (AF), control group (C) and placebo group (P), each containing 25 participants. The acupuncture points will be located and described according to the WHO Standard Acupuncture Locations. Based on the beneficial effects of previous clinical trials, the acupoints selected for this study will be: BL23, BL25, BL40, SP6 and KI3.

Interventions Participants of the LF, HF and AF groups will be submitted to the treatment protocol, which will consist of the bilateral application of electroacupuncture using a previously calibrated electrostimulator (Sikuro DS100C), consisted of alternating symmetrical biphasic waves with continuous pulse train for the low (2Hz) or high (100Hz) frequency groups, and a mixed pulse train for the alternating frequency group (100Hz and 2Hz for 3 seconds each); 100ms pulse duration and 0.5ms pulse width; and the maximum current (amplitude) intensity tolerated by the patient and intensified so that sensory habituation is avoided. Trichotomy will be carried out when necessary and the skin will be disinfected with 70% alcohol. With the participant lying down in a ventral position, the needles will be inserted at a 90º inclination with the skin, to a depth at which that the patient reports the "deQi" sensation (≅ 1.5cm).

The individuals that are randomly assigned to the C and P groups will follow exactly the same protocol as the electroacupuncture groups, however the C group will not undergo electrical stimulation, as the acupuncturist will activate channels that are not connected to the patient. In the P group an adhesive moxa (Dong Yang®) will be placed on each acupoint and the needle will be inserted over it, so that the participant only feels the needle prick, but without perforation of the skin and the "deQi" sensation. In addition, as in group C, the electrodes will be connected to the needles, however, no electrical current will be applied. Sterile and disposable 0.25mm x 30mm stainless steel needles (Dong Bang Acupuncture Inc., Seoul, Korea) will be used. The sessions will last 30 minutes, twice a week, for 5 weeks, totaling 10 sessions.

Sample size calculation The sample calculation was defined assuming a two-point difference in pain intensity through the Numerical Pain Scale, with an estimated standard deviation of 1.47 points. Considering a test power of 80%, a significance level of 5% and a sample loss of 20%, 25 participants will be recruited for each group (125 in total). (G * Power 3 3.1. 9.2).

Statistical analysis The statistical analysis will be performed according to the intention-to-treat principle. An analysis of variance (ANOVA) will be used to examine the effect of the treatment, time (pre- and post-treatment, 6 and 12 months follow up), and the interaction between groups versus time. If differences between the groups are identified, Tukey's multiple comparison test will be conducted. Two-sided paired t-tests will use for within-group comparisons (comparing baseline to follow up). The non-parametric statistical test (Kruskal Wallis) will be used if the data is not normally distributed. All statistical analyses will be conducted using SPSS (IBM Co, Armonk, New York, USA) for Windows, V.19.0. The confidence interval will be established at 95%, and the significance level will be set at 5%.

Safety At each treatment session the participants will be asked about any unpleasant and unintended signs or symptoms associated with the use of electroacupuncture. A questionnaire will also be used with a record of the duration and intensity of the adverse symptom reported by the patient, which will be scored according to a Likert-type scale from 1 to 5, with 1 representing the absence of adverse symptoms and 5 severe adverse symptoms.

Ethics and data security All the patients will participate voluntarily and will sign a consent form prior to the randomization. The access and storage of the data will be in accordance with the guidelines of the National Research Ethics Commission (CONEP). This study has been approved by the Ethics Committee of the University of São Paulo Medical School (authorization No. 2.903.991) and is registered in Plataforma Brasil (CAAE: 89846118.7.0000.0065).

ELIGIBILITY:
Inclusion Criteria:

* Over 60 years of age
* Either gender
* Diagnosis of nonspecific low back pain of more than 3 months duration, with or without radiating leg pain, with a minimum pain intensity score of 4 on the 11-point pain numerical rating scale (NRS - Brazilian Portuguese version)
* Walk independently (with or without walking devices)
* Agree to voluntarily participate in this study and sign the consent form.

Exclusion Criteria:

* Previous surgery on the spinal column
* Have a known or suspected serious spinal pathology (e.g., cancer, vertebral fracture, spinal infection or cauda equina syndrome)
* Fear of needles
* Have participated in acupuncture treatment in the previous 30 days
* Wheelchair users.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-12-18 (Estimated); Study Completion 2021-12-17 (Estimated)

PRIMARY OUTCOMES:
Pain intensity - Numerical Rating Scale (NRS) | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  Will be measure using the Numerical Rating Scale (NRS), an 11-point scale ranging from 0 (no pain) to 10 (worst possible pain). Participants will be asked to rate their average pain levels in the 24 hours prior to the assessment.
Pain intensity - Pressure pain threshold (PPT) | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  The PPT will be measured using a pressure algometer (EMG system, Brazil). The assessed region will be marked with a tape measure and a dermatographic pencil. Two points will be marked bilaterally: 5 cm to the right and left of the spinous process of L3 and L5. A control point will be marked on the anterior tibial muscle of the right leg, 5 cm lateral to the tuberosity of the tibia. The circular tip of the algometer will be positioned perpendicular to the participant's skin and gradually pressed until the participant reports that the pressure has become painful and unbearable. Three measurements will be taken at each point with an interval of 1 minute.

SECONDARY OUTCOMES:
Quality of pain | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  This will be analyzed using the McGill Pain Questionnaire, a valid and reliable instrument containing 78 pain descriptors divided into 4 categories (sensory, affective, evaluative and miscellaneous) and 20 subcategories, to which scores of 1 to 5 are attributed. The result is obtained by first scoring the words according to their position within the set of descriptors of each subcategory. The maximum score in the sensory category is 42, in the affective 14, in the evaluative 5 and in the miscellaneous 17. Then, the analysis is performed by adding these values associated with their categories. Higher scores equate to more intense pain.
Perceived overall effect | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  The patient's self-perception regarding the treatment will be evaluated using the Global Effect Perception Scale, a 11-point numerical scale ranging from -5 (much worse) to +5 (much better), where higher scores represent better recovery.
Emotional functionality - Depression | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  Depression will be assessed using the Beck Depression Inventory (BDI), a self-administered questionnaire that contains 21 items, with a score ranging from 0 to 3, where a higher score indicates more depressive symptoms.
Patient satisfaction | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  The evaluation of the patient's satisfaction with the treatment will be carried out using the MedRisk questionnaire of patient satisfaction with physiotherapeutic care. This questionnaire contains 20 items, covering global aspects of the treatment (2 items), aspects related to the service provided (8 items), and aspects about the therapist-patient relationship (10 items). Following a Likert-type scale, the patient's response will range from 1 (strongly disagree) to 5 (strongly agree), where higher scores represent greater satisfaction with the treatment.
Psychosocial factors | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  The risk of a poor prognosis due to psychosocial factors will be assessed using the STarT Back Screening Tool (SBST), a self-administered questionnaire with 9 items (4 related to referred pain and 5 related to psychosocial factors) where the patient has the response options "I agree" (1 point) and "I Disagree" (zero points) in the first eight items, and "Nothing", "A little" or "Moderate" (zero points each), "A lot" or "Extremely" (one point each) in the ninth item. If the total score is between 0-3 points, the patient is classified as low risk for poor prognosis. When the total score is greater than 3 points the score of the psychosocial subscale, questions 5 to 9, is then considered. If the score of this subscale is less than or equal to 3 points, the patient is classified as medium risk and scores greater than 3 points are considered to indicate a high risk for poor prognosis.
Physical functioning - Roland Morris Disability Questionnaire | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  This measure will be assessed through the Roland Morris Disability Questionnaire. This is a self-administered questionnaire, adapted to the Portuguese language, which aims to evaluate physical incapacity due to low back pain. This contains 24 items pertaining to activities that can be impaired due to LBP. Individuals need to select the items that apply to their pain on that day. The selected items are summed for a total score ranging from 0 to 24, with higher scores indicating more severe functional incapacity.
Emotional functionality - Anxiety | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  Anxiety will be assessed using the Global Anxiety - Visual Analog Scale (GA-VAS). This is composed of a 100mm line, where the left extremity is related to the absence of anxiety, and the right extremity is related to the worst possible anxiety. The individual is asked to assess the intensity of their anxiety in the previous 24 hours and to mark this on the line. The distance from the left edge of the line to the mark placed by the patient is measured in millimeters. Greater measurements indicate greater anxiety.
Physical functioning - Five Times Sit to Stand Test | prior to the start of treatment, immediately after the end of treatment (5 weeks), and at 6 and 12 months after the final treatment
  This measure will be assessed through the Five Times Sit to Stand Test (FTSST). The patient initiates the FTSST sitting in a chair without arm support, with the upper limbs crossed over the chest, feet positioned at hip width and knees in 90° flexion. They will be asked to stand and sit five times as fast as possible. A timer will be used to measure the task execution time. The test will be performed twice and the mean time will be calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Federal University of Parana, Curitiba, Paraná
  - University of Sao Paulo General Hospital, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within one year of study completion.
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Malta DC, Oliveira MM, Andrade SSCA, Caiaffa WT, Souza MFM, Bernal RTI. Factors associated with chronic back pain in adults in Brazil. Rev Saude Publica. 2017 Jun 1;51(suppl 1):9s. doi: 10.1590/S1518-8787.2017051000052. PMID 28591350
- [Background] Wong AYL, Karppinen J, Samartzis D. Low back pain in older adults: risk factors, management options and future directions. Scoliosis Spinal Disord. 2017 Apr 18;12:14. doi: 10.1186/s13013-017-0121-3. eCollection 2017. PMID 28435906
- [Background] Robinson HS, Dagfinrud H. Reliability and screening ability of the StarT Back screening tool in patients with low back pain in physiotherapy practice, a cohort study. BMC Musculoskelet Disord. 2017 May 31;18(1):232. doi: 10.1186/s12891-017-1553-x. PMID 28569152
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Chou R, Deyo R, Friedly J, Skelly A, Weimer M, Fu R, Dana T, Kraegel P, Griffin J, Grusing S. Systemic Pharmacologic Therapies for Low Back Pain: A Systematic Review for an American College of Physicians Clinical Practice Guideline. Ann Intern Med. 2017 Apr 4;166(7):480-492. doi: 10.7326/M16-2458. Epub 2017 Feb 14. PMID 28192790
- [Background] Langevin HM, Schnyer R, MacPherson H, Davis R, Harris RE, Napadow V, Wayne PM, Milley RJ, Lao L, Stener-Victorin E, Kong JT, Hammerschlag R; Executive Board of the Society for Acupuncture Research. Manual and electrical needle stimulation in acupuncture research: pitfalls and challenges of heterogeneity. J Altern Complement Med. 2015 Mar;21(3):113-28. doi: 10.1089/acm.2014.0186. Epub 2015 Feb 24. PMID 25710206
- [Background] Comachio J, Oliveira Magalhaes M, Nogueira Burke T, Vidal Ramos LA, Peixoto Leao Almeida G, Silva AP, Ferreira de Meneses SR, Costa-Frutuoso JR, Santos Miotto Amorim C, Pasqual Marques A. Efficacy of acupuncture and electroacupuncture in patients with nonspecific low back pain: study protocol for a randomized controlled trial. Trials. 2015 Oct 15;16:469. doi: 10.1186/s13063-015-0850-7. PMID 26472590
- [Background] Liu L, Skinner M, McDonough S, Mabire L, Baxter GD. Acupuncture for low back pain: an overview of systematic reviews. Evid Based Complement Alternat Med. 2015;2015:328196. doi: 10.1155/2015/328196. Epub 2015 Mar 4. PMID 25821485
- [Background] MacPherson H, Altman DG, Hammerschlag R, Youping L, Taixiang W, White A, Moher D; STRICTA Revision Group. Revised STandards for Reporting Interventions in Clinical Trials of Acupuncture (STRICTA): extending the CONSORT statement. PLoS Med. 2010 Jun 8;7(6):e1000261. doi: 10.1371/journal.pmed.1000261. PMID 20543992
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Nusbaum L, Natour J, Ferraz MB, Goldenberg J. Translation, adaptation and validation of the Roland-Morris questionnaire--Brazil Roland-Morris. Braz J Med Biol Res. 2001 Feb;34(2):203-10. doi: 10.1590/s0100-879x2001000200007. PMID 11175495
- [Background] Menezes Costa Lda C, Maher CG, McAuley JH, Hancock MJ, de Melo Oliveira W, Azevedo DC, Freitas Pozzi LM, Pereira AR, Costa LO. The Brazilian-Portuguese versions of the McGill Pain Questionnaire were reproducible, valid, and responsive in patients with musculoskeletal pain. J Clin Epidemiol. 2011 Aug;64(8):903-12. doi: 10.1016/j.jclinepi.2010.12.009. Epub 2011 Mar 27. PMID 21444194
- [Background] Gomes-Oliveira MH, Gorenstein C, Lotufo Neto F, Andrade LH, Wang YP. Validation of the Brazilian Portuguese version of the Beck Depression Inventory-II in a community sample. Braz J Psychiatry. 2012 Dec;34(4):389-94. doi: 10.1016/j.rbp.2012.03.005. PMID 23429809
- [Background] de Fatima Costa Oliveira N, Oliveira Pena Costa L, Nelson R, Maher CG, Beattie PF, de Bie R, Oliveira W, Camara Azevedo D, da Cunha Menezes Costa L. Measurement properties of the Brazilian Portuguese version of the MedRisk instrument for measuring patient satisfaction with physical therapy care. J Orthop Sports Phys Ther. 2014 Nov;44(11):879-89. doi: 10.2519/jospt.2014.5150. PMID 25361861
- [Background] Pilz B, Vasconcelos RA, Marcondes FB, Lodovichi SS, Mello W, Grossi DB. The Brazilian version of STarT Back Screening Tool - translation, cross-cultural adaptation and reliability. Braz J Phys Ther. 2014 Sep-Oct;18(5):453-61. doi: 10.1590/bjpt-rbf.2014.0028. Epub 2014 Aug 29. PMID 25372008
- [Background] Varoli FK, Pedrazzi V. Adapted version of the McGill Pain Questionnaire to Brazilian Portuguese. Braz Dent J. 2006;17(4):328-35. doi: 10.1590/s0103-64402006000400012. PMID 17262148
- [Background] Kahraman T, Ozcan Kahraman B, Salik Sengul Y, Kalemci O. Assessment of sit-to-stand movement in nonspecific low back pain: a comparison study for psychometric properties of field-based and laboratory-based methods. Int J Rehabil Res. 2016 Jun;39(2):165-70. doi: 10.1097/MRR.0000000000000164. PMID 27031182
- [Background] Gorenstein C, Andrade L, Vieira Filho AH, Tung TC, Artes R. Psychometric properties of the Portuguese version of the Beck Depression Inventory on Brazilian college students. J Clin Psychol. 1999 May;55(5):553-62. doi: 10.1002/(sici)1097-4679(199905)55:53.0.co;2-d. PMID 10392786
- [Background] Williams VS, Morlock RJ, Feltner D. Psychometric evaluation of a visual analog scale for the assessment of anxiety. Health Qual Life Outcomes. 2010 Jun 8;8:57. doi: 10.1186/1477-7525-8-57. PMID 20529361
- [Background] WHO standard acupuncture point locations in the Western Pacific Region. Manila, Philippines. 2009:1-242.
- [Background] Liu L, Skinner MA, McDonough SM, Baxter GD. Acupuncture for chronic low back pain: a randomized controlled feasibility trial comparing treatment session numbers. Clin Rehabil. 2017 Dec;31(12):1592-1603. doi: 10.1177/0269215517705690. Epub 2017 May 1. PMID 28459161
- [Background] Wang H, Yang G, Wang S, Zheng X, Zhang W, Li Y. The Most Commonly Treated Acupuncture Indications in the United States: A Cross-Sectional Study. Am J Chin Med. 2018 Oct 9:1-33. doi: 10.1142/S0192415X18500738. Online ahead of print. PMID 30298749
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708
- [Background] Yin C, Buchheit TE, Park JJ. Acupuncture for chronic pain: an update and critical overview. Curr Opin Anaesthesiol. 2017 Oct;30(5):583-592. doi: 10.1097/ACO.0000000000000501. PMID 28719458
- [Derived] Francescato Torres S, Brandt de Macedo AC, Dias Antunes M, Merllin Batista de Souza I, Dimitre Rodrigo Pereira Santos F, de Sousa do Espirito Santo A, Ribeiro Jacob F, Torres Cruz A, de Oliveira Januario P, Pasqual Marques A. Effects of electroacupuncture frequencies on chronic low back pain in older adults: triple-blind, 12-months protocol for a randomized controlled trial. Trials. 2019 Dec 23;20(1):762. doi: 10.1186/s13063-019-3813-6. PMID 31870456